CLINICAL TRIAL: NCT06895109
Title: Evaluation of Improvement in Cognitive Functions and Psychological Aspects in Patients With Severe Acquired Brain Injury After Cranioplasty
Brief Title: Cognitive Functions in Severe Acquired Brain Injury After Cranioplasty
Acronym: NeC
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, Direttore dell' Unità Operativa Complessa "Neuroriabilitazione ad alta intensità", Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6349
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Brain Injury; Neuropsychological Deficits; Cranioplasty; Cognitive Deficit Following Brain Lesions; Craniectomy; Brain Injury, Acute; Acquired Brain Injury; Rehabilitation; Rehabilitation Outcome; Cognitive Disorders; Neurorehabilitation
Keywords: brain injury; cranioplasty; cognitive deficit following brain lesions; neuropsychological deficits; craniectomy; neurosurgical procedure; neurorehabilitation; rehabilitation treatment; cognitive outcome; acquired brain injury; braininjury acute; craniocerebral injury
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary objective: The primary objective of the study is to analyze the neuropsychological profile of a sample of patients with severe acquired brain injury, who underwent craniotomy and subsequent opercular reapposition surgery 30 days after surgery.
  Interventions: Other: improvement of cognitive functions and psychological aspects
- Secondary objective: Evaluate the relationship between neuropsychological aspects and neurosurgical intervention of opercular re-opposition 7 days after surgery and any differences between 7 and 30 days; Analyze motor performance; Analyze cerebral metabolism of the patient sample. Analyze motor performance of the patient sample:
  Interventions: Other: improvement of cognitive functions and psychological aspects

INTERVENTIONS:
Other: improvement of cognitive functions and psychological aspects — To analyze the neuropsychological, motor and functional profile of a sample of patients with severe acquired brain injury, who underwent craniotomy and subsequent opercular reapposition surgery

SUMMARY:
Cranioplasty is the main reconstructive neurosurgical procedure, performed in approximately 80% of patients who have previously undergone demolitive surgeries in an emergency setting, particularly in the case of decompressive craniectomy . It mainly aims to ensure the protection of brain tissue and improve the aesthetic appearance. Statistical correlation analyses between timing of cranioplasty and neurological recovery are probably in favor of early cranioplasty. Cranioplasty improves motor and cognitive rehabilitation outcomes. However, it carries an increased risk of postoperative complications, such as seizures and infections. Other studies show that cranioplasty performed 3 to 6 months after craniectomy can significantly improve motor and cognitive recovery.

The timing of the intervention plays a fundamental role in enucleating cognitive improvement. In fact, greater cognitive changes have been observed in patients who underwent cranioplasty within 6 months of the injury. Therefore, cranioplasty must be considered a key factor for neuropsychological recovery and should be performed early in order to make the most of the rehabilitation window. In the literature, there are studies that have evaluated how cranioplasty can facilitate cognitive recovery, regardless of timing. In particular, a significant cognitive recovery was observed in the period immediately following cranioplasty, while the improvement stabilizes after a certain period of time and recovery begins to slow down. In patients with severe acquired brain injury (GCA), cranioplasty seems to significantly improve neuropsychological and motor function, even after a long time from the procedure. The aim of the study is therefore to evaluate whether in patients with severe acquired brain injury who underwent cranioplasty in the neurorehabilitation setting there is an improvement in cognitive, motor functions and psychological aspects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 to 79 years;

  * Patient with severe acquired brain injury, undergoing craniotomy and subsequent percolate repositioning;
  * Patient without cognitive disorders before GCA;
  * Patient with cognitive and/or psychological disorders post GCA;
  * Patient, caregiver or legal guardian, has voluntarily signed the informed consent, privacy form, approved by the Ethics Committee, before performing any procedure of the study

Exclusion Criteria:

* Age <18 or over 80;

  * An MMSE score less than 8;
  * Language barrier;
  * Education level less than 8 years of age (lower secondary school diploma);
  * Medical conditions such as severe hearing loss or vision loss that in the opinion of the physician could preclude data collection;
  * History of psychiatric disorders according to D5M V or ICD-10 criteria, for which, in the opinion of the physician, the patient is not suitable for enrollment;
  * Onset of acute pathologies close to the post-operative period and related to the surgery (1-10 days), such as: hydrocephalus, brain infections, epileptogenic picture.
  * Ongoing acute pathologies, liver, kidney or heart failure.
  * Patient, caregiver or legal guardian, refuse to sign the informed consent, privacy form, approved by the Ethics Committee, before performing any study procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with severe acquired brain injury who underwent craniotomy and subsequent opercular reapposition who met the inclusion criteria and did not meet any exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological profile | At baseline (T0) and 30 days after surgery (T1)
  To analyze the neuropsychological profile of a sample of patients with severe acquired brain injury, who underwent craniotomy and subsequent opercular reapposition surgery

SECONDARY OUTCOMES:
Analyze the various aspects | At T0: at the time of admission (pre-surgery); At T1: approximately one week after the operculum repositioning procedure; > At T2: approximately one month after the operculum repositioning procedure.
  To evaluate the relationship between neuropsychological aspects and neurosurgical intervention of opercular reopposition, to analyze motor performances, cerebral metabolism and motor performances of the patient sample.

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Neuroriabilitazione ad alta intensità, Fondazione Policlinico Universitario "A. Gemelli", Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheikh MA, Ali S, Khan A. Uroflowmetry: nomograms in healthy young Pakistani men. J Pak Med Assoc. 2024 Oct;74(10):1806-1810. doi: 10.47391/JPMA.10626. PMID 39407375
- [Background] Corallo F, Lo Buono V, Calabro RS, De Cola MC. Can Cranioplasty Be Considered a Tool to Improve Cognitive Recovery Following Traumatic Brain Injury? A 5-Years Retrospective Study. J Clin Med. 2021 Nov 21;10(22):5437. doi: 10.3390/jcm10225437. PMID 34830718
- [Background] Corallo F, Calabro RS, Leo A, Bramanti P. Can cranioplasty be effective in improving cognitive and motor function in patients with chronic disorders of consciousness? A case report. Turk Neurosurg. 2015;25(1):193-6. doi: 10.5137/1019-5149.JTN.10618-14.2. PMID 25640571
- [Background] Di Stefano C, Rinaldesi ML, Quinquinio C, Ridolfi C, Vallasciani M, Sturiale C, Piperno R. Neuropsychological changes and cranioplasty: A group analysis. Brain Inj. 2016;30(2):164-71. doi: 10.3109/02699052.2015.1090013. Epub 2015 Dec 8. PMID 26647093
- [Background] De Cola MC, Corallo F, Pria D, Lo Buono V, Calabro RS. Timing for cranioplasty to improve neurological outcome: A systematic review. Brain Behav. 2018 Nov;8(11):e01106. doi: 10.1002/brb3.1106. Epub 2018 Oct 2. PMID 30280509
- [Background] Malcolm JG, Rindler RS, Chu JK, Grossberg JA, Pradilla G, Ahmad FU. Complications following cranioplasty and relationship to timing: A systematic review and meta-analysis. J Clin Neurosci. 2016 Nov;33:39-51. doi: 10.1016/j.jocn.2016.04.017. Epub 2016 Aug 4. PMID 27499122
- [Background] Corallo F, De Cola MC, Lo Buono V, Marra A, De Luca R, Trinchera A, Bramanti P, Calabro RS. Early vs late cranioplasty: what is better? Int J Neurosci. 2017 Aug;127(8):688-693. doi: 10.1080/00207454.2016.1235045. Epub 2016 Sep 28. PMID 27609482
- [Background] Ozoner B. Cranioplasty Following Severe Traumatic Brain Injury: Role in Neurorecovery. Curr Neurol Neurosci Rep. 2021 Oct 21;21(11):62. doi: 10.1007/s11910-021-01147-6. PMID 34674047
- [Background] Corallo F, De Cola MC, Lo Buono V, Cammaroto S, Marra A, Manuli A, Calabro RS. Recovery of Severe Aphasia After Cranioplasty: Considerations on a Case Study. Rehabil Nurs. 2020 Jul/Aug;45(4):238-242. doi: 10.1097/rnj.0000000000000212. PMID 30681549